CLINICAL TRIAL: NCT03798925
Title: Microbiological Diagnostic Performance of Metagenomic Next-generation Sequencing for Pulmonary Infection in Clinical Settings
Brief Title: mNGS for Detection of Pathogens for Pulmonary Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Department of Infectious Diseases, Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-mNGS-respiratory
Record Dates: First submitted 2018-12-29; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None Intervention — It is observational study

SUMMARY:
Pulmonary infections remain the leading causes of morbidity and mortality among patients worldwide. Pathogen identification is crucial yet difficult for the majority of the cases. Metagenomic Next-generation Sequencing provides a potential technology for rapid and untargeted pathogen detection for pulmonary infection. The study is designed observationally to investigate if mNGS is superior to traditional paradigm of serial tests in the aspect of diagnostic performance. Patients whose primary diagnosis is pulmonary infetion and bronchoalveolar lavage fluid can be obtained will be enrolled. Both mNGS and traditional paradigm of serial tests wil be performed.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary infection as the primary diagnosis
* Bronchoalveolar lavage fluid can be obtained

Exclusion Criteria:

* when the primary diagnosis is tumor or connective tissue diseases
* microbiological diagnosis is confirmed before bronchoalveolar lavage
* not enough bronchoalveolar lavage fluid for mNGS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients whose primary diagnosis is pulmonary infetion and bronchoalveolar lavage fluid can be obtained
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-19 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
microbiological diagnosis (pathogen of pulmonary infection) | through study completion, up to 6 months
  the final microbiological diagnosis (pathogen of pulmonary infection) after using of every detection method and combined with clinical manifestations.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided